CLINICAL TRIAL: NCT00625222
Title: Transcranial Direct Current Stimulation (tDCS) As A Tool For Prospective Responder Identification Before Vagus Nerve Stimulation (VNS) Implantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Luebeck (Other)
Collaborators: Cyberonics, Inc. (Industry); University Hospital, Bonn (Other); University of Erlangen-Nürnberg Medical School (Other); Epilepsycenter Bielefeld (Unknown)
Responsible Party: Prof. Jürgen Sperner, M.D., Pediatrics Department, University of Luebeck, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: tDCS-VNS001; AZ07-135
Record Dates: First submitted 2008-02-11; First posted 2008-02-28 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2010-01

CONDITIONS: Epilepsy
Keywords: Electroencephalography; Seizure frequency; Seizure severity
MeSH Terms: conditions — Epilepsy | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: transcranial direct current stimulation

INTERVENTIONS:
Procedure: transcranial direct current stimulation — 1mA, 15 Minutes, constant direct current

SUMMARY:
The aim of the study is to establish tDCS as a prognostic tool to predict VNS therapy outcome among patients with pharmacoresistant epilepsy.

DETAILED DESCRIPTION:
In recent years it has been shown that many different brain stimulation techniques are effective in seizure reduction in epilepsy patients as well as in animal models of epilepsy. VNS is the method most often used with at least 45.000 patients implanted with this device worldwide. However, prediction of seizure outcome after VNS implantation is not possible in an individual patient so far. Recently, tDCS is increasingly used as a method to reduce seizure frequency in epileptic patients. Therefore it is hypothesized, that a positive effect after a single tDCS, in terms of short time seizure reduction and reduction of epileptic discharges in the EEG, could be predictive for epilepsy outcome after VNS implantation.

In the proposed multicenter prognostic study we test the predictive value of tDCS for each patient with refractory epilepsy 1 week up to 2 months before VNS implantation. The effects of tDCS will be verified via a 15 minutes long routine EEG examination, performed immediately before and after tDCS, together with seizure diary and seizure severity scale, assessed 1 month before and 1 week after tDCS. A 6 months long observation period will follow the VNS implantation. At the end of the 6 months period seizure diary and seizure severity scale of the last month will be performed to measure VNS therapy outcome. On the basis of the described variables, immediate up to 1 week long tDCS effects will be correlated to 6 months long VNS therapy outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age: 12 years and above
* At least 2 years disease history
* Refractory epilepsy:

  * Seizures are not completely responsive to longlasting antiepileptic treatment. At least 4 antiepileptic medicaments failed in mono or combined anticonvulsive regimen.
  * At least 4 seizures per week in the last month, despite adequate antiepileptic regimen.
  * Epilepsy surgery is not indicated or not accepted by the patient or by the parents of the patient.
* A stable anticonvulsive regimen, defined as unchanged dose and type of the antiepileptic medication in the last month before tDCS and before VNS implantation.
* Seizure diary is available and completed.
* VNS implantation is planned within the next 2 months.

Exclusion Criteria:

* Acute, symptomatic seizures (caused by tumor, stroke, acute encephalitis)
* Uncontrolled medical problems (e.g. cardiovascular, nephrotic oder severe, chronic or severe acute disease)
* Increased intracranial pressure for whatever reason
* Implantation of metallic material (e.g. pacemaker, cochlear-implant)
* Diseased or damaged skin over the scalp (e.g. Dermatitis)
* Pregnancy
* Known or supposed non-compliance
* Age: less than 12 years

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Correlation of tDCS effects in terms of EEG changes, number of seizures and seizure severity to VNS therapy outcome | 6 Months

SECONDARY OUTCOMES:
To define criteria which will have predictive value for VNS therapy outcome. | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Sperner, Prof., M.D., Study Chair — Pediatrics Department, University of Luebeck, Germany; Iren Orosz, M.D., Principal Investigator — Pediatrics Department, University of Luebeck, Germany
Locations (1):
- Pediatrics Department, University of Luebeck, Lübeck, Germany